CLINICAL TRIAL: NCT07143240
Title: Tedizolid Neuropathies
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 25-5138
Record Dates: First submitted 2025-08-08; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Adult Patients Developing Optic or Peripheral Neuropathy; While Receiving Tedizolid Therapy Between July 2019 and December 2024
Keywords: Infectiology; tedizolid
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Adult patients developing optic or peripheral neuropathy while receiving tedizolid therapy: The study population included subjects aged ≥ 18 years who received tedizolid for infections between July 2019 and December 2024.
  Subjects younger than 18 years old were excluded.
  Interventions: Other: Determine patient demographic and clinical characteristics at baseline

INTERVENTIONS:
Other: Determine patient demographic and clinical characteristics at baseline — Description of demographic data (sex, age), comorbidities (Charlson scores), septic history, clinical data relating to neuropathy, and tedizolid prescription modalities (dose, duration).

SUMMARY:
Tedizolid is a new oxazolidinone, related to linezolid. It has obtained marketing authorization for the treatment of skin and soft tissue infections. Its potential interest compared to linezolid lies mainly in its better tolerance in the context of more prolonged treatments required in chronic Gram-positive cocci infections such as osteoarticular infections. Indeed, linezolid has hematological toxicity, appearing beyond 10 days of treatment. Due to a lower dosage and lower mitochondrial toxicity, the hematological tolerance of tedizolid is better, even allowing it to be used as a relay from linezolid after the occurrence of hematotoxicity. Another side effect of the oxazolidinone class is the occurrence of optic and peripheral neuropathies observed under linezolid. The pharmacological properties of tedizolid and in vitro and in vivo data suggested a lower risk of neurotoxicity, although a few cases have been published..

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* Patients developing optic or peripheral neuropathy while receiving tedizolid therapy

Exclusion Criteria:

* 18 years

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients developing optic or peripheral neuropathy while receiving tedizolid treatment.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Describe cases of tedizolid-induced neurotoxicity. | The outcome will be measured at the last follow-up visit in 2024, i.e. a maximum of 4 years after the start of the neuropathy.
  Retrospective cohort describing neurological side effects occurring under tedizolid. Patients will be identified by cross-referencing data from medical records of the infectious diseases department of the Lyon University Hospital, the prospective database of CRIOAc Lyon recording the side effects of new molecules (including tedizolid), and pharmacovigilance data. Description of patient history and clinical data, and tedizolid prescription methods (dose, duration).
  Unit of Measure :Number of patients (n)

CONTACTS AND LOCATIONS:
Locations (1):
- HCL, Lyon, France, France